CLINICAL TRIAL: NCT00661011
Title: A Phase II Study Assessing the Curative Effect of the Combination of Lobectomy Followed by Mediastinal Concomitant Radiochemotherapy in Patients With Locally Advanced Unresectable Stage III Non-small Cell Lung Cancer Responding to Induction Chemotherapy
Brief Title: Lobectomy and Mediastinal Radiochemotherapy in Unresectable Stage III Non-Small Cell Lung Cancer Responding to Induction Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to too slow recruitment
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELCWP 01061
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non-small cell lung carcinoma; Concomitant radiochemotherapy; Cisplatin; Vinorelbine; Radiotherapy; Chemotherapy; Unresectable stage III non-small cell lung carcinoma; Surgery; Unresectable stage III non-small cell lung carcinoma not suitable for radical radiotherapy after objective response to induction chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Lobectomy followed by mediastinal concomitant chemoradiotherapy
  Interventions: Procedure: Lobectomy followed by concomitant mediastinal chemoradiotherapy

INTERVENTIONS:
Procedure: Lobectomy followed by concomitant mediastinal chemoradiotherapy — Lobectomy Radiotherapy 66 Gy in 2 Gy/ fraction, 5 fractions/wk Chemotherapy Cisplatin 60 mg/m² on days 1 and 22 and Vinorelbine 15 mg/m² on days 1, 8, 22 and 29

SUMMARY:
The purpose of this study is to determine if radical radiochemotherapy on the mediastinum after lobectomy can be associated with significant long term survival in patients with initially unresectable stage III NSCLC responding to induction chemotherapy but in which the residual disease is too large to be treated by radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell carcinoma of the lung
* Initially stage III NSCLC
* Pathologically proven N2 or N3 disease
* Any response to induction chemotherapy (whatever the regimen administered)
* Disease still not fully resectable (because of extensive mediastinal N disease) and not suitable for radical radiotherapy (single field) after induction chemotherapy
* Lobectomy possible for the treatment of T disease
* Availability for participating in the detailed follow-up of the protocol
* Informed consent

Exclusion Criteria:

* Prior treatment with radiotherapy or surgery
* Karnofsky PS < 60
* Functional or anatomical contra-indication to mediastinal radiotherapy
* Functional or anatomical contra-indication to surgical lobectomy
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or cured malignant tumour (more than 5 year disease-free interval)
* Malignant pleural or pericardial effusion
* Neutrophils < 2,000/mm³
* Platelet cells < 100,000/mm3
* Serum bilirubin > 1.5 mg/100 ml
* Serum creatinine > 1.5 mg/100 ml and/or creatinine clearance < 60 ml/min
* Recent myocardial infarction (less than 3 months prior to date of diagnosis)
* Congestive cardiac failure or cardiac arrhythmia requiring medical treatment
* Uncontrolled infectious disease
* Hearing loss
* Symptomatic polyneuropathy
* Serious medical or psychological factors which may prevent adherence to the treatment schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Survival | Survival will be dated from the day of registration until death or last follow up

SECONDARY OUTCOMES:
Operative mortality and morbidity | To be observed during the 30 days following the surgical procedure
Local control rate | After completion of treatment
Toxicity | After each course of chemotherapy and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Sculier, MD, PhD, Study Chair — European Lung Cancer Working Party
Locations (12):
- Belgium (10):
  - Department of Pneumology RHMS Hôpital de la Madeleine, Ath
  - Department of Pneumology CHR St Joseph-Warquignies, Boussu
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology Hospital Ixelles-Molière, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Hôpital Vésale - Montigny-le-Tilleul, Montigny-le-Tilleul
  - Department of Pneumology Centre Hospitalier de Mouscron, Mouscron
  - CH Peltzer-La Tourelle, Verviers
- Medical Oncology St Savas Hospital, Athens, Greece
- Medical Oncology Hospital de Sagunto, Valencia, Spain

REFERENCES:
- See also: (Click here for more information on the protocol) — http://www.elcwp.org